CLINICAL TRIAL: NCT02187016
Title: A Randomized, Parallel Design Study to Assess the Effects of Three Interproximal Cleaning Modalities Versus a Manual Toothbrush Control on Gingivitis and Plaque Following a Period of Home Use
Brief Title: Efficacy and Safety Study of Interproximal Cleaning Modalities on Oral Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philips Oral Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MAH-13-0151
Record Dates: First submitted 2014-07-01; First posted 2014-07-10 (Estimated); Results first posted 2015-12-29 (Estimated); Last update posted 2016-03-08 (Estimated); Status verified 2016-02

CONDITIONS: Gingivitis
Keywords: Gingivitis; plaque; interproximal cleaning; dental floss
MeSH Terms: conditions — Gingivitis; Plaque, Amyloid | interventions — Dental Devices, Home Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- AirFloss + BreathRx (Experimental): Device: Subjects brushed with a ADA Reference Manual Toothbrush once a day for 1 minute. Subjects used interproximal cleaning device with BreathRx rinse once a day.
  Interventions: Device: AirFloss + BreathRx
- AirFloss + Listerine (Experimental): Device: Subjects brushed with a ADA Reference Manual Toothbrush once a day for 1 minute. Subjects used interproximal cleaning device with Listerine Cool Mint rinse once a day.
  Interventions: Device: AirFloss + Listerine
- Dental Floss (Experimental): Device: Subjects brushed with a ADA Reference Manual Toothbrush once a day for 1 minute. Subjects used interproximal cleaning device once a day.
  Interventions: Device: Dental Floss
- Manual Toothbrush (Active Comparator): Device: Subjects brushed with a ADA Reference Manual Toothbrush once a day for 1 minute
  Interventions: Device: Manual Toothbrush

INTERVENTIONS:
Device: AirFloss + BreathRx — Manual Toothbrush used twice daily, 1 minute. Interproximal cleaning plus Rinse used once daily.
  Arms: AirFloss + BreathRx
Device: AirFloss + Listerine — Manual Toothbrush used twice daily, 1 minute. Interproximal cleaning plus Rinse used once daily.
  Arms: AirFloss + Listerine
Device: Dental Floss — Manual Toothbrush used twice daily, 1 minute. Interproximal cleaning used once daily.
  Arms: Dental Floss
Device: Manual Toothbrush — Manual Toothbrush used twice daily, 1 minute.
  Arms: Manual Toothbrush

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of tooth and interproximal cleaning modalities with and without chemistry on oral health over 28 days.

ELIGIBILITY:
Inclusion Criteria:

* Be willing and physically able to carry out all study procedures and be available at all times required for participation
* Be able to fully understand and comply with the written and verbal instructions provided
* Provide written Informed Consent
* Be age 18 - 65 years
* Agree to return study materials at the required visits
* Be a non-smoker
* Have a minimum of 20 'scorable' teeth (excluding 3rd molars)
* Have a minimum average plaque score of > 0.5 per RMNPI scoring with 2-6 hours of plaque accumulation
* Have a Gingival Bleeding Index of ->1 on at least 10 sites
* Be a regular manual toothbrush user
* Be a non or irregular flosser defined as using dental floss or any other interproximal cleaning technique once per week or less often

Exclusion Criteria:

* A medical or dental condition that would be unduly affected by participation in this study, per Investigator discretion
* Pregnant or nursing per subject report
* A medical condition requiring antibiotic pre-medication prior to dental appointments
* Diagnosis of xerostomia
* Any oral or extra oral piercing that interferes with the ability to perform study procedures and/or clinical assessments in the mouth
* Currently undergoing or requiring dental/periodontal treatment, or having had periodontal treatment in the six months preceding the study, where the subject's study participation could present an undue safety risk or obscure the evaluation of study endpoints, per Investigator /Examiner discretion
* Oral surgery within the last 2 months
* Current use of professionally dispensed bleaching products
* A known allergy or sensitivity to products planned for use in this study
* Unwillingness to abstain from all other oral hygiene products other than those prescribed for the duration of the study
* Unwillingness to abstain from all other oral hygiene products other than those prescribed for the duration of the study
* Participation in an oral care study within the previous 90 days
* Be an employee or a relative of an employee of the Site clinical research department, dental school, or a dental products manufacturing, research or marketing firm
* Are a dental student or dental professional
* A cardiac pacemaker or implanted cardiac defibrillator
* Insulin-Dependent Diabetes
* Current use of antibiotic medications or use within 4 weeks of enrollment
* Current use of prescription-dose anti-inflammatory medications or anticoagulants; (including aspirin > 81 mg daily)
* Presence of advanced periodontal disease or excessive gingival recession, per Investigator/Examiner discretion
* Heavy deposits of calculus, either supragingival and/or subgingival, per Investigator/Examiner discretion
* Extensive crown or bridge work and/or rampant decay, per Investigator/Examiner discretion
* Presence of orthodontic bands interfering with efficacy outcome(s) per Investigator/Examiner discretion
* Have a professional prophylaxis within 4 weeks of the study
* Be a regular power toothbrush user

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 290 (Actual)
Dates: Start 2014-06; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pejmon Amini, DDS, Principal Investigator — Silverston Research Group
Locations (1):
- Silverstone Research Group, Las Vegas, Nevada, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- AirFloss + Rinse1: AirFloss interproximal cleaning device with BreathRx applied once a day between the teeth with Manual Tooth brushing twice a day for 1 minute.
- AirFloss + Rinse2: AirFloss interproximal cleaning device with Listerine applied once a day between the teeth with Manual Tooth brushing twice a day for 1 minute.
- String Floss: String Floss interproximal cleaning device is applied once a day between the teeth with Manual Tooth brushing twice a day for 1 minute
- Manual Toothbrush: Manual Toothbrush is used twice a day for 1 minute
Period: Overall Study
Arm/Group | AirFloss + Rinse1 | AirFloss + Rinse2 | String Floss | Manual Toothbrush
Started | 80 | 80 | 79 | 51
Completed | 79 | 78 | 78 | 51
Not Completed | 1 | 2 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AirFloss + Rinse1 | AirFloss + Rinse2 | String Floss | Manual Toothbrush | Total
Number analyzed (Participants) | 79 | 78 | 79 | 51 | 287
Age, Continuous [Mean (Standard Deviation); unit: years] | 37 (12.20) | 35.6 (10.70) | 34.9 (11.00) | 35.1 (12.10) | 35.7 (11.50)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 50 | 51 | 33 | 184
  Male | 29 | 28 | 28 | 18 | 103
Region of Enrollment [Number; unit: participants]
  United States | 79 | 78 | 79 | 51 | 287

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Gingival Inflammation on a 4 Point Scale Using the Modified Gingival Index (MGI) at Day 14
Description: MGI is a validated assessment of Gingival inflammation using a 4 point range where 0 (absence of inflammation) to 4 (severe inflammation).
Time Frame: 14 days
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | AirFloss + Rinse1 | AirFloss + Rinse2 | String Floss | Manual Toothbrush
Number analyzed (Participants) | 79 | 78 | 79 | 51
units on a scale | 0.10 (0.01) | 0.10 (0.01) | 0.10 (0.01) | 0.01 (0.01)

2. Secondary Outcome: Change From Baseline in Gingival Inflammation on a 4 Point Scale Using the Modified Gingival Index (MGI) at Day 28
Description: MGI is a validated assessment of Gingival inflammation using a 4 point scale from 0 (absence of inflammation) to 4 (severe inflammation).
Time Frame: 28 days
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | AirFloss + Rinse1 | AirFloss + Rinse2 | String Floss | Manual Toothbrush
Number analyzed (Participants) | 79 | 78 | 78 | 51
units on a scale | 0.20 (0.01) | 0.22 (0.01) | 0.26 (0.01) | 0.03 (0.02)

3. Secondary Outcome: Change From Baseline in Gingival Bleeding Index (GBI) on a 4 Point Scale at Day 14
Description: GBI is a validated assessment of gingival bleeding using a 4 point scale with 0 (no bleeding) to 3 (spontaneous bleeding).
Time Frame: 14 days
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | AirFloss + Rinse1 | AirFloss + Rinse2 | String Floss | Manual Toothbrush
Number analyzed (Participants) | 79 | 78 | 79 | 51
units on a scale | 0.05 (0.00) | 0.05 (0.00) | 0.05 (0.00) | 0.00 (0.01)

4. Secondary Outcome: Change From Baseline in Gingival Bleeding Index (GBI) on a 4 Point Scale at Day 28
Description: as for outcome 3
Time Frame: 28 days
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | AirFloss + Rinse1 | AirFloss + Rinse2 | String Floss | Manual Toothbrush
Number analyzed (Participants) | 79 | 78 | 78 | 51
units on a scale | 0.08 (0.00) | 0.08 (0.00) | 0.09 (0.00) | 0.01 (0.01)

5. Secondary Outcome: Change From Baseline Using Rustogi Modification of the Navy Plaque Index (RMNPI) Using a Dichotomous Scale at Day 14
Description: RMNPI is a validated assessment of visual surface dental plaque using a dichotomous scale 0 (absence) to 1 (presence).
Time Frame: 14 days
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | AirFloss + Rinse1 | AirFloss + Rinse2 | String Floss | Manual Toothbrush
Number analyzed (Participants) | 79 | 78 | 79 | 51
units on a scale | 0.09 (0.01) | 0.10 (0.01) | 0.11 (0.01) | 0.04 (0.01)

6. Secondary Outcome: Change From Baseline in Rustogi Modification of Navy Plaque Index (RMNPI) Using a Dichotomous Scale at Day 28
Description: RMNPI is a validated assessment of visual surface dental plaque using a dichotomous scale 0 (absence) to 1 (presence).
Time Frame: 28 days
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | AirFloss + Rinse1 | AirFloss + Rinse2 | String Floss | Manual Toothbrush
Number analyzed (Participants) | 79 | 78 | 78 | 51
units on a scale | 0.15 (0.01) | 0.16 (0.01) | 0.17 (0.01) | 0.04 (0.01)

ADVERSE EVENTS:
Time Frame: Oral changes from baseline evaluated at Day 14 and 28
Arm/Group | AirFloss + Rinse1 | AirFloss + Rinse2 | String Floss | Manual Toothbrush
Serious Adverse Events (participants affected / at risk) | 0/79 | 0/78 | 0/78 | 0/51
Other Adverse Events (participants affected / at risk) | 2/79 | 1/78 | 1/78 | 0/51
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AirFloss + Rinse1 (N=79) | AirFloss + Rinse2 (N=78) | String Floss (N=78) | Manual Toothbrush (N=51)
Gingival Irritation (Injury, poisoning and procedural complications) | 2 | 1 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No